CLINICAL TRIAL: NCT04274985
Title: Reliability, Validity of The Turkish Version of Fonseca Anamnestic Index
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Halime ARIKAN, Research Assistant, Gazi University
Other Study IDs: 91610558-604.01.02-
Record Dates: First submitted 2020-02-16; First posted 2020-02-18 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2022-01

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Validity; Reliability; Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1: Patients with temporomandibular disorders
  Interventions: Other: Questionnaire application

INTERVENTIONS:
Other: Questionnaire application — Patients will complete the mentioned questionnaires.

SUMMARY:
The aim in this study is to determine the Turkish version validity and reliability of the Fonseca Anamnestic Index.

DETAILED DESCRIPTION:
Approximately 60% of individuals with temporomandibular disorders (TMD) reported increased pain intensity from midlevel to severe. This was seen at the end of the intervention or work related activities in the quarter of individuals. Therefore, the correct diagnosis of TMD is very important to reduce the economic cost. Fonseca Anamnestic Index (FAI) is an easy and understandable questionnaire. This questionnaire consists of 10 questions that provide a versatile evaluation of the temporomandibular joint (TMJ) in the head and neck, whether there is pain during chewing, the presence of parafunctional habits, range of motion, joint sounds, malocclusion, and emotional stresses. The participants give one of the answers to the questions "Yes = 10 points, Sometimes = 5 points, No = 0 points". As a result of the total of the points, the participants are evaluated as "TMD-None = 0-15 points, Mild-TMD = 20-40 points, Moderate TMD = 45-60 points, Severe-TMD = 100 points". The aim of this study was to evaluate the validity and reliability of the Turkish version of FAI. The study of validity and reliability is planned with 50 individuals with TMD. The sociodemographic characteristics of the individuals will be questioned by the investigators and then the patients will be evaluated with FAI, Craniofacial Pain and Disability Inventory (CF-PDI), Neck Disability Index (NDI), Tampa Scale for Kinesiophobia (TSK), Pain Catastrophizing Scale (PCS), Headache Impact Test-6 (HIT-6), Jaw Functional Limitation Scale (JFLS) (Turkish version) and Visual Analogue Scale (VAS). The test-retest will be re-administered by face-to-face interview technique after 1 week. The results will be analyzed using the SPSS version 22.0 computer package program.

ELIGIBILITY:
Inclusion Criteria:

* Having a temporomandibular disorder
* Individuals who suited Temporomandibular Disorders/ Research Diagnostic Criteria classification

Exclusion Criteria:

* Pregnant,
* Canser,
* Trauma,
* Neurologic disorder,
* Infection,
* Trigeminal or postherpatic neuralgia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with temporomandibular disorders between the ages of 18-50
Sampling Method: Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Fonseca Anamnestic Index (FAI) | 5 minutes
  Fonseca Anamnestic Index (FAI) is an easy and understandable questionnaire. This questionnaire consists of 10 questions that provide a versatile evaluation of the temporomandibular joint (TMJ) in the head and neck, whether there is pain during chewing, the presence of parafunctional habits, range of motion, joint sounds, malocclusion, and emotional stresses. The participants give one of the answers to the questions "Yes = 10 points, Sometimes = 5 points, No = 0 points". As a result of the total of the points, the participants are evaluated as "TMD-None = 0-15 points, Mild-TMD = 20-40 points, Moderate TMD = 45-60 points, Severe-TMD = 100 points".It is valid and reliable a questionnaire in clinic. Therefore, Turkish version must do.

CONTACTS AND LOCATIONS:
Locations (1):
- Halime ARIKAN, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Derived] Arikan H, Citaker S, Ucok C. Psychometric properties of the Fonseca Anamnestic Index (FAI) for temporomandibular disorders: Turkish version, responsiveness, reliability, and validity study. Disabil Rehabil. 2024 Apr;46(7):1408-1415. doi: 10.1080/09638288.2023.2199221. Epub 2023 Apr 17. PMID 37066863